CLINICAL TRIAL: NCT05119192
Title: Dual-Tasking for Individuals With Lower Limb Amputation: Exploring the Relationship to Falls and Instrumental Activities of Daily Living
Acronym: DIAL
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: VA Eastern Colorado Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: A3640-M; RX003640-01A1 (Other Grant/Funding Number: Veterans Administration RR&D)
Record Dates: First submitted 2021-11-01; First posted 2021-11-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Amputation
Keywords: Dual-task; Falls; Activities of Daily Living; Lower-limb amputation; Avascular Amputation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — no biospecimen retention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Veterans with Dysvascular Lower Limb Amputation: Self-report assessments, performance-based assessments, and optional individual interview with Veterans with dysvascular lower limb amputation.

SUMMARY:
Veterans with dysvascular lower limb amputation (LLA) have a high fall risk, which persists despite completion of conventional rehabilitation. The presence of fall risk could be a primary reason for the high disability and low quality of life outcomes in this Veteran population. A potential novel intervention for this population is to train performance of tasks that require both physical and cognitive attention (i.e., dual-tasking). Therefore, the purpose of this study is to explore relationships between dual-task performance and self-reported falls for Veterans with dysvascular LLA. Further, dual-tasking occurs during everyday life and this project will examine the association between dual-task performance and participation in activities of daily living (basic and instrumental). The results will form the foundation for development and future study of a novel dual-task training program for Veterans with dysvascular LLA.

DETAILED DESCRIPTION:
Purpose: To explore the relationship between dual-task performance, self-reported falls, and activities of daily living for Veterans with lower limb amputation.

Dual-task performance will be assessed using overground ambulation and serial subtraction. Dual-tasking will then be compared to single-task silent walking or seated serial subtraction to determine the category each participant falls into: gait-priority trade off, cognitive-priority trade off, mutual facilitation, or mutual interference. Self-reported falls with be assessed with questionnaires including recent falls (1 month, 1 year), number of falls, fall injuries, and near-falls. Activities of daily living will be assessed using the Modified Barthel Index, and Frenchay Activities Index. Other self-report descriptive questionnaires include: demographic information, the Functional Comorbidities Index, and the Falls Behavioral Scale for the Older Person. Other performance measures include: the Berg Balance Scale, and the SLUMS cognitive screen.

Aim 1: Compare the proportion of participants experiencing mutual interference during dual-task walking between fall groups (Non-fall is 1 fall vs. Recurrent-fall is >1 fall).

Aim 2: Identify the relationships dual-task effects have with self-reported participation in activities of daily living (basic and instrumental ADLs).

Aim 3: Qualitatively explore the effects of dual-tasking on self-reported fall or near-fall dual-task scenarios. Veterans with dysvascular LLA (n 30) will participate in semi-structured interviews describing these scenarios, and dual-task awareness in fall prevention.

ELIGIBILITY:
Inclusion Criteria:

* unilateral, transtibial, or transfemoral LLA
* diagnosis of diabetes mellitus or peripheral artery disease
* age 50 to 89 years
* able to ambulate around the home with or without an assistive device
* at least one year since LLA

Exclusion Criteria:

* trauma or cancer-related etiology of the LLA
* decisionally challenged individuals (SLUMS score in "Dementia" range)
* prisoners
* active cancer treatment
* clinical discretion of principle investigator to exclude patients who are determined to be unsafe and/or inappropriate to participate in the described intervention

Ages: 50 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Veterans with dysvascular lower-limb amputation
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Dual-task Performance | Baseline
  Dual-task performance will be classified into one of 4 categories (gait priority trade off, cognitive priority trade off, mutual interference, or mutual facilitation) based on performance in 3 different 2-minute conditions (gait single task, cognitive single task, dual-task). The gait task will be overground walking on a 12 meter obstacle-free course with a 1 meter turning area. Gait speed (m/s) will be calculated using the total distance covered over the 2 minutes. The cognitive task will be serial subtractions of seven, starting between 590-599. A corrected response rate will be calculated as: responses per second*percent of correct responses. Dual-task performance will represent a participant's performance on improvement or decline on both gait and cognitive performance comparing single and dual-tasking. For example, mutual interference would be a decline in both gait (slower speed), and cognitive (lower corrected response ratio) from single to dual-tasking.

SECONDARY OUTCOMES:
Self-reported falls | Baseline
  Participants will be asked: "How many times have you fallen in the last year?". Participants will be provided with the definition of a fall as: "an unexpected event in which.[you] come to rest on the ground, floor, or lower level" excluding intentional change in position. To account for potential disproportion of Fall groups, follow-up questions will be asked, including: near-falls in the past year, and presence of fear of falling.
Modified Barthel Index | Baseline
  The Modified Barthel Index assesses 10 different ADLs, with the overall score ranging from 0 (total dependence) to 100 (independence). The MBI has been used effectively for individuals with dysvascular LLA one year after amputation, and demonstrates excellent test-retest reliability in the outpatient setting.
Frenchay Activities Index | Baseline
  The Frenchay Activities Index is pragmatic for community-dwelling adults to self-rate participation in three domains: domestic chores, leisure/work, and outdoor activities. Frenchay Activity Index scores range from 15-60, with higher scores indicating greater participation in instrumental ADLs.

CONTACTS AND LOCATIONS:
Overall Officials: Laura A. Swink, PhD, Principal Investigator — Rocky Mountain Regional VA Medical Center, Aurora, CO
Locations (1):
- Rocky Mountain Regional VA Medical Center, Aurora, CO, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
When results are published a final de-identified, anonymized data set may be made available to the public, based on availability of resources for the given journal publisher. Care will be taken to ensure that individuals cannot be re-identified in the dataset, with no inclusion of or links to personally identifiable information.

DOCUMENTS (1):
  • Informed Consent Form (2022-03-15): https://cdn.clinicaltrials.gov/large-docs/92/NCT05119192/ICF_000.pdf